CLINICAL TRIAL: NCT03318614
Title: Bifidobacterium Infantis M-63 Improves Mental Health in Irritable Bowel Syndrome Developed After a Major Flood Disaster
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Morinaga Milk Industry Co., LTD (Industry)
Responsible Party: Principal Investigator, Yeong Yeh Lee, Professor Dr, Universiti Sains Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/15040133
Record Dates: First submitted 2017-10-12; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Irritable Bowel Syndrome; Abdominal Pain; Small Intestinal Bacterial Overgrowth
Keywords: Gut Microbiota; Probiotics; Abdominal Pain; Small Intestinal Bacterial Overgrowth; Mental
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants assigned to the M-63 group were given a sachet of B. infantis M63 (2.5 x 109 cfu/g per sachet) (Morinaga Milk Industry Co. Ltd., Japan) to consume daily for three months in addition to advice of good hygiene and sanitation practices. No drug intervention was given to the control group over three months other than advice of good hygiene and sanitation practices.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics M-63 group (Experimental): Participants assigned to the M-63 group were given a sachet of B. infantis M63 (Morinaga Milk Industry Co., Ltd., Japan) to consume daily in addition to advice of good hygiene and sanitation practices.
  Interventions: Dietary Supplement: Probiotics M-63
- Control group (Placebo Comparator): No probiotic intervention was given to the control group over three months other than advice of good hygiene and sanitation practices.
  Interventions: Other: Control group

INTERVENTIONS:
Dietary Supplement: Probiotics M-63 — B. infantis M63 (2.5 x 109 cfu/g per sachet) was given to Probiotics M-63 group for three months.
  Arms: Probiotics M-63 group
Other: Control group — No probiotic intervention was given to the control group for three months.
  Arms: Control group

SUMMARY:
A 3-month study was conducted in flood victims from affected villages in the Tumpat district, Kelantan. Participants were given either probiotic, Bifidobacterium infantis M63 (M-63 group) or no probiotics (control group) for three months. At baseline and 3-month, participants were assessed for thewater, sanitation and hygiene (WaSH) practices, abdominal symptoms, breath testing for hydrogen and methane to detect the presence of SIBO and also fecal samples for gut microbiota profiling.

DETAILED DESCRIPTION:
There is an observed rise in cases of acute gastroenteritis and post-infectious irritable bowel syndrome (PI-IBS) during the peak flood period. One major reason is poor sanitation, water and hygiene practice by flood victims during the flood because of poor access to clean water. The mechanism how poor hygiene causes non-specific abdominal complaints is unknown. The investigators speculated that small intestinal overgrowth (SIBO) is the fundamental basis for the increase in reported cases of acute gastroenteritis and abdominal complaints among flood victims. The investigators further speculated that administration of antibiotics or probiotics could reduce the abdominal symptoms after three months.

Therefore, the intervention study was conducted for three months. Compliance of participants was checked by a diary given to participants in the M-63 group to document their daily intake of probiotics. This study will for the first time demonstrate the fundamental mechanism behind the poor WaSH practices and gastrointestinal disturbances after flood. Also this study would support a role for probiotic intervention to reduce abdominal complications when the next flood occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years; flood victims who fulfilled the Rome III criteria for IBS developed after flood, able to perform breath-testing, able to provide stool specimens, and able to complete three months of prospective intervention.

Exclusion Criteria:

* Adults who took antibiotics or probiotics three months prior to and after flood had taken place; previous abdominal surgery and presence of significant medical and psychiatric co-morbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
IBS Symptom Severity Scale (IBS-SSS) scores | Three months
  IBS-SSS contains five questions that determine severity of abdominal pain, severity of abdominal distension, dissatisfaction with bowel habits and interference with quality of life (QOL) on a 100-point visual analogue scale. Since each question contributes to the score equally, therefore 500 is the maximum score, and higher the score, the severity is worse. For those participants with scores below 175, they have mild IBS, and in general, if scores are below 75, they are considered in remission. No units of measure are used.

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36) scores | Three months
  SF-36 measures four physical components (i.e. physical functioning, role limitations in physical health, bodily pain and general health perception) and four mental components (i.e. social functioning, role limitations due to emotional problems, vitality or energy and mental well-being). Total physical component and total mental component were calculated as the sum of all items in the physical and mental components, respectively. Participants with a higher score in each domain of SF-36 have a better quality of life (QOL) in that domain. No units of measure are used.
Hospital Anxiety and Depression Scale (HADS) scores | Three months
  The Malay-translated version of 14-item HADS contains four-point Likert responses Participants with higher scores had worse anxiety and depression. No units of measure are used.
Breath-testing for small intestinal bacterial overgrowth (SIBO) | Three months
  Participants were asked to exhale end-expiratory breath samples into a collection bag at baseline. Then they were asked to drink 75 g of glucose in cold water. At intervals of 15 mins for the next 2 hours, breath samples were collected and symptoms recorded. Forty mL of exhaled breath were syringed into the machine (Quintron, Milwaukee, US), and levels of H2 and CH4 (in parts per million or ppm) were determined. For a positive test, the following criteria were applied: a rise in H2 value (≥ 20 ppm) or CH4 values (≥ 10 ppm) above fasting baseline value or a sustained rise in H2 or CH4 of 5 ppm over 3 consecutive breath samples. A rise in breath values as above and reproduction of symptoms were required to diagnose SIBO.
Changes in gut microbiota at the phylum level | Three months
  Fresh fecal specimens were collected and gut microbial analysis was performed. Changes in gut microbiota at the phylum level were reported in terms of relative abundance.

CONTACTS AND LOCATIONS:
Overall Officials: Yeong Yeh Lee, MD, PhD, Principal Investigator — Universiti Sains Malaysia

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Ma ZF, Yusof N, Hamid N, Lawenko RM, Mohammad WMZW, Liong MT, Sugahara H, Odamaki T, Xiao J, Lee YY. Bifidobacterium infantis M-63 improves mental health in victims with irritable bowel syndrome developed after a major flood disaster. Benef Microbes. 2019 Mar 13;10(2):111-120. doi: 10.3920/BM2018.0008. Epub 2018 Dec 10. PMID 30525951